CLINICAL TRIAL: NCT06213714
Title: The 5th Generation Tele-Robotic-Assisted Percutaneous Coronary Intervention: A First-in-Human Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yan'an Affiliated Hospital of Kunming Medical University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Kunming Chenggong District People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5G Tele-Robotic-Assisted PCI
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Cardiovascular Diseases; Coronary Disease; Arteriosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Cardiovascular Diseases; Coronary Disease; Arteriosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5G Tele-Robotic-Assisted PCI (Experimental): VRS100 Robotic Console System, was developed by Shenzhen Raysight Intelligent Medical Technology Co., Ltd., will be used for 5G Tele-Robotic-Assisted Percutaneous Coronary Intervention in this study.
  Interventions: Device: 5G Tele-Robotic-Assisted PCI

INTERVENTIONS:
Device: 5G Tele-Robotic-Assisted PCI — The 5G Tele-Robotic-Assisted VRS100 system is intended for use in the remote delivery and manipulation of guidewires and rapid exchange balloon/stent catheters, and remote manipulation of guide catheters during percutaneous coronary intervention (PCI) procedures.
  Other Names: VRS100 Robotic Console System

SUMMARY:
The objective of this study is to examine the safety and effectiveness, from both clinical and technical perspectives, of utilizing the 5G-Robotic VRS100 system in percutaneous coronary intervention (PCI).

ELIGIBILITY:
Inclusion Criteria:

* General Inclusion Criteria:

  1. Age ≥18 years.
  2. Patients with coronary artery disease undergoing Percutaneous Coronary Intervention (PCI).
  3. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.
* Angiographic Inclusion Criteria:

  1. De-novo coronary artery disease.
  2. Reference vessel diameter is 2.5-4.0mm by visual estimate.
  3. Target lesion length is ≤30.0mm.
  4. Target lesion is a single de-novo native coronary artery lesion. This lesion may consist of multiple lesions (with ≤10mm between diseased segments) and must be completely covered by a single stent with ≥5.0mm of normal segments on proximal and distal edges of the lesion.
  5. Target lesion diameter showing stenosis ≥70% by visual estimate, or ≥50% with myocardial ischemia.
  6. Target lesion angiography meets the calculation criteria of Rui-Xin AngioQFA, and AngioQFA is ≤0.8.

Exclusion Criteria:

* Patients meeting any of the following criteria will be excluded:
* General Exclusion Criteria:

  1. Subjects with indications for urgent PCI surgery.
  2. Evidence of an acute myocardial infarction within one week prior to the intended VRS100 procedure.
  3. Subject has undergone PCI within 72 hours prior to the VRS100 procedure.
  4. Subject has undergone PCI within 30 days prior to the VRS100 procedure and experienced a MACE or a serious adverse event (SAE).
  5. Severe heart failure (NYHA IV & LVEF≤35%).
  6. Subject has suffered a stroke, or has an active peptic ulcer or upper gastrointestinal bleeding within 6 months prior to planned VRS100 procedure.
  7. Subject has known hypersensitivity or contraindication to aspirin, heparin, ticagrelor, clopidogrel, bivalirudin, PTX(paclitaxel), stainless steel, etc.
  8. Subject has acute or chronic kidney disease (serum creatinine level of >2.5 mg/dL or >221 umol/L) or need dialysis.
  9. Pregnant or breastfeeding, or planning to be pregnant.
  10. Repeated enrollment.
  11. Any other factors that the researchers consider not suitable for inclusion or completion of this study.
* Angiographic Exclusion Criteria:

  1. Any previous stent placement within 5.0 mm (proximal or distal) of the target lesion.
  2. Target lesion requires planned treatment with directional coronary atherectomy (DCA), laser, rotational atherectomy or any device except for balloon dilatation prior to stent placement.
  3. Cardiac allograft vasculopathy (CAV).
  4. Target lesion/vessel has evidence of intraluminal thrombus.
  5. Chronic total occlusion (CTO).
  6. Target lesion located in a native vessel distal to an ostial, bifurcation or anastomosis.
  7. Unprotected left main coronary artery disease defined as an obstruction greater than 50% diameter stenosis in the left main coronary artery.
  8. Target lesion or vessel proximal to the target lesion has severe tortuosity or calcification.
  9. Target lesion that cannot be fully covered by a single stent.
  10. More than 2 lesions requires treatment in one vessel.
  11. Subject requires treatment of more than one vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 48 hours or hospital discharge, whichever occurs first
  Defined as angiographic success (residual stenosis after stenting of <30% with final TIMI [Thrombolysis In Myocardial Infarction] flow grade 3) without an in-hospital major adverse cardiovascular event (MACE) (cardiovascular death, MI, clinically driven target vessel revascularization).
Technical Success | 1 day
  Defined as the successful advancement and retraction of PCI devices using the VRS100 System and without conversion to manual operation.

SECONDARY OUTCOMES:
PCI Procedure Time | During procedure
  Defined as the time measured from the insertion of the guide catheter until the removal of the guide catheter.
Overall Procedure Time | During procedure
  Defined as the time measured from the insertion of the hemostasis sheath until the removal of the guide catheter.
Fluoroscopy and/or X-Ray Time | During procedure
  As recorded by an X-Ray System utilized during the procedure.
Patient Radiation Exposure - Cumulative Dose | During procedure
  Cumulative dose (mGy) as recored during the procedure.
Contrast Fluid Volume | During procedure
  The amount of contrast fluid used (mL) during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Study Chair — Shanghai Zhongshan Hospital; Chenguang Li, Principal Investigator — Shanghai Zhongshan Hospital; Qiang Xue, Principal Investigator — Yan'an Affiliated Hospital of Kunming Medical University; Wangxiong Li, Principal Investigator — Kunming Chenggong District People's Hospital

IPD SHARING:
Plan to Share IPD: No